CLINICAL TRIAL: NCT02433054
Title: Bern Venous Stent Registry
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Nils Kucher, Professor, University of Zurich
Other Study IDs: 262/ 2014
Record Dates: First submitted 2015-03-27; First posted 2015-05-04 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Post-thrombotic Syndrome
Keywords: deep vein thrombosis; chronic venous disease; May-Thurner syndrome; venous stent
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis; May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (1):
- CE-certified dedicated venous stents: Patients receiving self-expanding venous nitinol stents.
  Interventions: Device: CE-certified dedicated venous stents

INTERVENTIONS:
Device: CE-certified dedicated venous stents — Implantation of self-expanding nitinol venous stents in the iliofemoral veins and/or inferior vena cava.

SUMMARY:
The purpose of this study is to examine patency rates of self-expanding nitinol stents for treatment of iliofemoral and inferior vena cava residual thrombosis, obstruction or stenosis. Moreover, clinical outcome data of patients treated with these venous stents will be collected.

DETAILED DESCRIPTION:
Background: Obstruction and stenosis of the ilio-femoro-caval veins are difficult to treat by conservative measures only. Despite anticoagulation and consequent use of compression stockings, lower extremity venous hypertension affects patients quality of life and health status by causing venous claudication, swelling, skin changes, and venous ulcers. In the last decades venous stenting has become an accepted treatment for ilio-femoro-caval obstruction. Recently, novel self-expanding nitinol stents have been specifically designed for the venous system to account for the anatomical structure of ilio-femoro-caval veins.

Gap of Knowledge: There are few data on short and long term outcomes of self-expanding Nitinol stent placement in ilio-femoro-caval veins.

Objective: To study patency rates and clinical outcome data of self-expanding Nitinol stents that were specifically designed for iliofemoral and inferior vena cava residual thrombosis, obstruction or stenosis.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving self-expanding venous nitinol stents for one of the following indications:

* Residual thrombosis of iliofemoral veins and/or inferior vena cava after thrombus removal (by catheter-directed thrombolysis or pharmacomechanical thrombolysis)
* Post-thrombotic syndrome and chronic obstruction of iliofemoral veins and/or inferior vena cava
* Chronic venous insufficiency and presence of non-thrombotic venous stenosis of iliofemoral veins and/or inferior vena cava

Exclusion Criteria:

* No consent
* Inability to provide informed consent
* Allergy to Nitinol
* Pregnancy, breast-feeding or birth-giving during the last 30 days
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of chronic venous disease and obstruction and/or stenosis of the iliofemoral veins and/or inferior vena cava.
Sampling Method: Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Primary patency rate | after one year up to a follow-up of five years

SECONDARY OUTCOMES:
Primary assisted patency rate | after one year up to a follow-up of five years
Target vessel revascularization | after one year up to a follow-up of five years
Secondary patency rate | after one year up to a follow-up of five years
Revised Venous Clinical Severity Score | after one year up to a follow-up of five years
CEAP-Score | after one year up to a follow-up of five years
Adverse events: Stent-related: Rethrombosis (early and late), In-Stent restenosis, Stent compression/fracture Clinical: Postthrombotic syndrome, Bleeding (major, minor), Death (VTE-related, Bleeding-related, other), Recurrent VTE at any site | after one year up to a follow-up of five years

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof. Dr. med., Principal Investigator — University Hospital Zurich, Clinic of Angiology
Locations (1):
- Klinik für Angiologie, Universitätsspital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Sebastian T, Barco S, Kreuzpointner R, Konstantinides S, Kucher N. Reversal of cardiopulmonary exercise intolerance in patients with post-thrombotic obstruction of the inferior vena cava. Thromb Res. 2021 Dec;208:219-225. doi: 10.1016/j.thromres.2021.03.025. Epub 2021 Apr 9. PMID 33840477
- [Derived] Sebastian T, Gnanapiragasam S, Spirk D, Engelberger RP, Moeri L, Lodigiani C, Kreuzpointner R, Barco S, Kucher N. Self-Expandable Nitinol Stents for the Treatment of Nonmalignant Deep Venous Obstruction. Circ Cardiovasc Interv. 2020 Dec;13(12):e009673. doi: 10.1161/CIRCINTERVENTIONS.120.009673. Epub 2020 Dec 4. PMID 33272030
- [Derived] Sebastian T, Spirk D, Engelberger RP, Dopheide JF, Baumann FA, Barco S, Spescha R, Leeger C, Kucher N. Incidence of Stent Thrombosis after Endovascular Treatment of Iliofemoral or Caval Veins in Patients with the Postthrombotic Syndrome. Thromb Haemost. 2019 Dec;119(12):2064-2073. doi: 10.1055/s-0039-1697955. Epub 2019 Oct 28. PMID 31659739
- [Derived] Sebastian T, Engelberger RP, Spirk D, Hakki LO, Baumann FA, Spescha RS, Kucher N. Cessation of anticoagulation therapy following endovascular thrombus removal and stent placement for acute iliofemoral deep vein thrombosis. Vasa. 2019 Jul;48(4):331-339. doi: 10.1024/0301-1526/a000774. Epub 2019 Jan 22. PMID 30667348
- [Derived] Sebastian T, Hakki LO, Spirk D, Baumann FA, Periard D, Banyai M, Spescha RS, Kucher N, Engelberger RP. Rivaroxaban or vitamin-K antagonists following early endovascular thrombus removal and stent placement for acute iliofemoral deep vein thrombosis. Thromb Res. 2018 Dec;172:86-93. doi: 10.1016/j.thromres.2018.10.027. Epub 2018 Oct 26. PMID 30391776
- [Derived] Sebastian T, Dopheide JF, Engelberger RP, Spirk D, Kucher N. Outcomes of endovascular reconstruction of the inferior vena cava with self-expanding nitinol stents. J Vasc Surg Venous Lymphat Disord. 2018 May;6(3):312-320. doi: 10.1016/j.jvsv.2017.11.012. Epub 2018 Mar 15. PMID 29550177